CLINICAL TRIAL: NCT00938444
Title: Prospective, Multicenter, Non-interventional Study in RA Patients Treated With Tocilizumab - Evaluation of the BRADA and ABILHAND Questionnaires
Brief Title: Evaluation of the BRADA and ABILHAND Questionnaires
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Filip De Keyser, MD PhD, University Hospital Ghent
Other Study IDs: 2009/190; ML22613
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Patients with moderate to severe RA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with moderate to severe RA: Patients with moderate to severe RA treated with Tocilizumab

SUMMARY:
This protocol is designed to evaluate the BRADA and ABILHAND questionnaires in rheumatoid arthritis (RA) patients that will be treated with an effective therapy. Patients with moderate to severe RA treated with tocilizumab will be asked to complete the BRADA and ABILHAND questionnaires at screening, baseline, after 12 weeks and after 24 weeks of treatment. All other assessments and questionnaires from daily clinical practice (such as the global assessment of disease activity by the patient, the Health Assessment Questionnaire (HAQ), the SF36 questionnaire, measurement of ESR and CRP and the DAS 28 calculation), will also be used to evaluate these questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* patients with moderate to severe RA.
* Inadequate response on earlier optimal use of a minimum of two DMARDs (disease modifying anti-rheumatic drugs such as goldsalts, salazopyrine, leflunomide, methotrexate (MTX)) as far as one of the two used DMARDs is MTX that at the exception of a documented intolerance despite the association with folic acid, should have been administered IM or oral during a minimum of 3 months and at a minimal dose of 15mg/week.
* DAS 28 score ≥ 5.1
* For whom a drug that is registered for the treatment of moderate to severe RA is commercially available but does not constitute a satisfactory treatment for this patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe RA.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the BRADA and ABILHAND questionnaires to detect clinically important changes over time. | after 24 weeks of treatment with tocilizumab

CONTACTS AND LOCATIONS:
Overall Officials: Filip De Keyser, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (19):
- Belgium (19):
  - Jan Palfijn, Merksem, Antwerpen
  - ASZ, Aalst
  - Clinique St. Luc, Bouge
  - CHU Brugmann, Brussels
  - UCL St. Luc, Brussels
  - UZA, Edegem
  - AZ Sint-Lucas, Ghent
  - University Hospital Ghent, Ghent
  - Reuma Instituut, Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Gasthuisberg, Leuven
  - CHU de Liège, Liège
  - CH Notre Dame - R Fabiola, Montignies-sur-Sambre
  - Clinique St. Pierre, Ottignies
  - Clinique St. Vincent, Rocourt
  - Heilig Hartziekenhuis, Roeselare
  - AZ Alma, Sijsele
  - Hôpital de Jolimont, Soignies
  - UCL Mont-Godinne, Yvoir

REFERENCES:
- [Derived] Janssens X, Decuman S, De Keyser F; Brada I study group. Construction and psychometric properties of the Belgian Rheumatoid Arthritis Disability Assessment (BRADA) questionnaire: a new tool for the evaluation of activity limitations in patients with rheumatoid arthritis. Clin Exp Rheumatol. 2013 Jul-Aug;31(4):596-605. Epub 2013 Jul 30. PMID 23899969
- See also: website of the University Hospital Ghent — http://www.uzgent.be